CLINICAL TRIAL: NCT05871385
Title: rTMS Plus Vestibular Rehabilitation as an Adjunct Treatment for Fall Risk and Postural Instability for Chronic Vestibular Dizziness Patients, Double Blinded RCT
Brief Title: rTMS Plus Vestibular Rehabilitation as an Adjunct Treatment for Fall Risk and Postural Instability for Chronic Vestibular Dizziness Patients/ Chronic Labyrinthitis
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samir Abdelkhalik Youssef, lecturer at faculty of physical therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002202
Record Dates: First submitted 2023-04-22; First posted 2023-05-23 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Vestibular Disorders
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (r TMS group) (Experimental): Twenty eight randomly assigned patients with peripheral vestibular disorders will undergo 10 Hz rTMS to the dorsolateral prefrontal cortex of their dominant hemisphere; in addition to designed vestibular rehabilitation exercises.
  Device: repetitive transcranial magnetic stimulation high frequency (10 HZ) rTMS pulses are applied to the dorsolateral prefrontal cortex of the dominant hemisphere.
  Interventions: Device: rTMS group
- Control (Group B) (placebo rTMS) (Placebo Comparator): Twenty eight randomly assigned patients with peripheral vestibular disorders will undergo placebo rTMS plus designed vestibular rehabilitation exercises.
  Interventions: Device: placebo rTMS group

INTERVENTIONS:
Device: rTMS group — Twenty eight randomly assigned patients with peripheral vestibular disorders will undergo 10 Hz rTMS to the dorsolateral prefrontal cortex of their dominant hemisphere; in addition to designed vestibular rehabilitation exercises
  Other Names: repetitive transcranial magnetic stimulation
  Arms: Group A (r TMS group)
Device: placebo rTMS group — Twenty eight randomly assigned patients with peripheral vestibular disorders will undergo placebo rTMS plus designed vestibular rehabilitation exercises.
  Other Names: placebo rTMS
  Arms: Control (Group B) (placebo rTMS)

SUMMARY:
Falling is one of the most common consequences of vestibular dizziness. Most of patients with vestibular dysfunction suffer from balance disorders, postural instability and vertigo that may lead to life threating complications as fractures and brain injuries. Non invasive brain stimulation techniques such as repetitive transcranial magnetic stimulation (rTMS) have been investigated as therapeutic interventions for various neurological disorders like motor deficits and balance disorders after various neurological deficits. To investigate the effect of repetitive transcranial magnetic stimulation (rTMS) added to supervised vestibular rehabilitation program on balance and postural stability in patients with vestibular dizziness

DETAILED DESCRIPTION:
The subjects of both genders with age 40 to 65 will be allocated randomly into two equal groups A and B. Group A Outcomes measure will include : Berg balance scale, computerized dynamic posturography (CDP) . Assessment will be done before and after treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with peripheral vestibular disorders from audiologist or neurologist.
2. The patient's age will be ranged from forty five to seventy years old.
3. Patients will experience at least two symptoms of common symptoms of peripheral vestibular disorders.
4. Symptoms of vertigo and nystagmus lasting from seconds to one minute.
5. Vertigo that arises from changes in head position related to gravity.
6. Patients who experienced symptoms for more than three months (chronic patients)
7. Patients were selected to be ambulant.
8. Patients suffer from balance disturbance with low risk falling (41-56) and moderate risk falling ranges (21-40) according to berg balance scale.
9. All patients were medically stable, controlled with medical drugs for at least three months and failed to medical treatment with no other physical, mental or cognitive disorders.

Exclusion Criteria:

1. Central vestibular disorders ( Ms, ataxia, migraine headache, posterior inferior cerebellar artery syndrome "PICA").
2. Vertigo that arises from changes in head position not related to gravity; as vertigo of cervical origin or vascular origin ( Vertebro- basilar insufficiency "VBI").
3. Previous surgery of the ear.
4. Bilateral peripheral vestibular weakness, central vestibular weakness, mixed vestibular weakness, or acute vestibular weakness.
5. Unstable health issues (cardiac dysfunction, end stage renal failure, unstable diabetes, uncontrolled hypertension >190/110…).
6. Pacemaker or other implanted electrically sensitive device.
7. Significant orthopedic or chronic pain syndrome (e.g any condition that wouldn't permit to completion of any of the tests).
8. Major cognitive dysfunction. neurodegenerative disease or major psychiatric condition ( Alzheimer's disease , depression….).
9. Chronic use of medications that could influence motor or sensory excitability (e.g AEDs, antipsychotic).
10. Alcohol abuse.
11. Epilepsy.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Postural stability | change from baseline to 8 weeks after intervention
  Computerized dynamic Posturography- Scores ranging zero min score and 100 max score
Visual Vertigo Analogue Scale | change from baseline to 8 weeks after intervention
  Indicate the amount of dizziness you experience in different situations

SECONDARY OUTCOMES:
Berg balance scale | change from baseline to 8 weeks after intervention
  Balance
  * 14 items each item scored from zero (min score)-4 (Max score) with total min score zero and max score 56

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University Hospitals, Cairo
  - faculty of medicine , Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided